CLINICAL TRIAL: NCT00430599
Title: The Effect of Levetiracetam (Keppra) on the Treatment of Tremor in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3384
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
We are carrying out this study to determine whether Keppra (a drug usually used to treat epilepsy) is an effective treatment for tremor in patients with Multiple Sclerosis. Tremor is one of the most common symptoms in MS, but also one of the most difficult to treat. A very small previous study has indicated that Keppra may be effective in this role, but we need to reproduce these results in many more patients before we can reliably confirm this.

DETAILED DESCRIPTION:
Multiple Sclerosis is the most common inflammatory demyelinating disease of the CNS and is the leading cause of neurological disability in young adults in the UK (~ 90,000 patients' affected). It has been estimated that the direct cost to the National Health Service is over £300 million/year and the total cost to UK society exceeds £1.3 billion/year. The personal cost in terms of disability is also high with 50% of patients requiring aids to walk or being wheelchair bound within 16 years of disease onset. Recently, attention has focused on disease modifying drugs, including b-Interferon, which have demonstrated a significant reduction in clinical relapse rate associated with a dramatic reduction in disease activity on brain MRI4-7. However, the evidence for any sustained long term benefit is poor. Therefore, symptomatic therapies remain a key part of patient management.

Cerebellar tremor and cerebellar gait instability are present in up to 70% of chronic MS patients and account for a significant amount of clinical morbidity. Cerebellar tremor is a major therapeutic problem in MS since currently there are no effective treatments. To date medical therapies including propranolol, clonazepam, carbamazepine, isoniazid, phenobarbitone, ondansetron, topiramate, gabapentin and cannabis have all been studied with little sustained benefit. More radical surgical treatments including thalamotomy and Deep Brain Stimulation have also been attempted.

However, a recent pilot study, with a small number of patients, suggested that Keppra (Levetiracetam) is effective in treating MS tremor. This study relied upon a rather subjective assessment of tremor and did not assess patients using quantitative physiological measures.

This protocol involves a collaboration between a clinical neurologist, with a recognised expertise in MS, and a research group with an established expertise in the electrophysiological and pharmacological investigation of human tremor11. The protocol describes a study, in MS patients, designed to establish whether Keppra (Levetiracetam) produces:

1. Physiologically measurable reduction in tremor;
2. Subjective and qualitative reduction in tremor;

ELIGIBILITY:
Inclusion Criteria:

1. McDonald criteria for diagnosis of MS (McDonald, 2001)15
2. Clinical evidence of Cerebellar Tremor.
3. Aged 18-60

Exclusion Criteria:

1. There is evidence of a further significant MS relapse during the trial
2. Evidence of resting tremor, or Holmes (rubral) tremor
3. Pregnant or breast feeding mothers
4. Patients with inadequate understanding of the English language to comprehend the patient information sheet
5. Evidence of any significant renal impairment
6. History of epilepsy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with multiple sclerosis and clinical evidence of cerebellar tremor.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-02; Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr P Nichols, MRCP, DPhil, Principal Investigator — Newcastle NHS Hospitals Trust
Locations (1):
- Sir James Spence Institute, Royal Victoria Infirmary, Newcastle, Tyne and Wear, United Kingdom